CLINICAL TRIAL: NCT02159144
Title: Cold Stress Stimulate the Browing of Subcutaneous White Adipose in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xiang Guang-da (Other)
Responsible Party: Sponsor-Investigator, Xiang Guang-da, Director of Endocrinology Department, Wuhan General Hospital of Guangzhou Military Command
Organization: Wuhan General Hospital of Guangzhou Military Command (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2014Wze088
Record Dates: First submitted 2014-05-31; First posted 2014-06-09 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Obesity; Type 2 Diabetes
Keywords: Brown adipose tissue; Subcutaneous white adipose tissue; White adipose tissue
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — Cold-Shock Response

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- healthy adults (Experimental)
  Interventions: Other: cold stress

INTERVENTIONS:
Other: cold stress

SUMMARY:
Adipose tissues, which include white adipose tissue (WAT) and brown adipose tissue (BAT), play an essential role in regulating whole-body energy homeostasis. Recent studies also reveal the presence of a subset of cells in WAT that could be induced by environmental or hormonal factors to become ''brown-like'' cells, and this ''beigeing'' process has been suggested to have strong antiobesity and antidiabetic benefits. More recently, same studies showed that cold stress stimulate the browning of subcutaneous white adipose. However, to the investigators knowledge, there are no direct data that clearly show that cold stress can promote the browning of subcutaneous white adipose.

DETAILED DESCRIPTION:
Individuals have cold exposure at 15C for 2 hr everyday for one week.Biopsy for subcutaneous white adipose was performed before and after one week cold exposure programme under local anesthesia. Measure the brown fat characteristics of biopsy samples. The expression levels of uncoupling protein-1 (UCP-1), peroxisome proliferator-activated receptor (PPAR)-r, peroxisome proliferator-activated receptor r coactivator 1 a (PGC1a) , growth factor receptor binding protein-10 (Grb10), PR domain containing 16 (PRDM16) will be determined before and after cold stress programme from the biopsy samples. In addition, a combination of PET and computed tomography (CT) - with the glucose analogue 18F-fluorodeoxyglucose (18F-FDG) as a tracer will be performed for brown adipose tissue before and after cold stress programme.

ELIGIBILITY:
Inclusion Criteria:

* healthy men
* 18-60 years old
* BMI 20-28 kg/m2

Exclusion Criteria:

* BMI < 20 kg/m2
* BMI > 28 KG/M2
* Female

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
browning of subcutaneous white adipose | 4 months
  Brown fat characteristics of biopsy samples will be assessed by determining the expression levels of UCP1, PGC1a, PRDM16 and Grb10.

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan General Hospital, Wuhan, Hubei, China